CLINICAL TRIAL: NCT06662695
Title: Effect of Oral Supplementation of Ginger on Plasma Cholesterol Efflux Capacity From THP-1 Macrophage
Brief Title: Ginger and Plasma Cholesterol Efflux Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Associate professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 43008844
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Ginger; HDL; cholesterol efflux; ABCA1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ginger (Experimental): Ginger-based supplement
  Interventions: Dietary Supplement: Ginger-based supplement
- Placebo (Placebo Comparator): Capsules containing corn flour
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ginger-based supplement — Ginger-based supplement in a dosage of 1500 mg
  Arms: Ginger
Dietary Supplement: Placebo — Capsules containing corn flour
  Arms: Placebo

SUMMARY:
In light of the findings from experimental studies examining the effects of ginger-derived compounds on cholesterol efflux pathways, this study aims to investigate the impact of oral ginger supplementation on high-density lipoprotein (HDL) function. The crossover and double-blind study will be conducted in two four-week periods, with a minimum of three weeks between these two phases. In one of the two study periods, participants will receive a ginger supplement, while in the other period, they will receive a placebo in the form of capsules. At the outset and end of each study period, venous blood samples will be obtained from the subjects. Plasma and buffy coat (containing white blood cells) will be separated and stored at -80. Cholesterol efflux capacity (CEC) will be determined by adding participants' plasma samples to the culture medium of THP-1 cells. Additionally, the gene expression of ATP-binding cassette transporters (ABCA1) and ABCG1 will be determined in the tissue lining obtained from the blood samples of the participants.

DETAILED DESCRIPTION:
The relationship between serum high-density lipoprotein cholesterol (HDL-C) and atherosclerosis was initially elucidated by the Framingham study. However, current evidence suggests that maintaining an optimal HDL-C level may not be sufficient to reduce the risk of cardiovascular disease (CVD). The majority of clinical trials have demonstrated that plasma HDL-C-raising drugs do not confer a reduction in the risk of developing CVD. Consequently, there has been a decline in interest in pursuing the elevation of HDL-C levels as a therapeutic objective. Mendelian randomization studies have called into question the causal relationship between plasma HDL-C levels and CVD. This may be due to factors related to HDL function and the reverse cholesterol transport pathway, including the effect of CEC. A number of studies involving large clinical populations have observed a robust inverse correlation between CEC and CVD after adjustment for plasma HDL-C levels. This suggests that CEC may serve as a more reliable biomarker for CVD than plasma HDL-C concentration. The efflux of cholesterol from macrophages may contribute to anti-inflammatory and anti-atherogenic effects, as well as reducing the accumulation of cholesterol esters in macrophages, which in turn leads to the production of foam cells. It is possible that ginger may affect this process. A limited number of in vitro studies have investigated the impact of ginger compounds on CEC, with all studies demonstrating a positive influence on the mediator of the reverse cholesterol transport pathway. These findings are in alignment with the results of an animal study in which hamsters fed a high-fat diet and ginger extract exhibited enhanced CEC. Moreover, it is conceivable that inflammatory processes may impede the efflux of cholesterol and the reverse cholesterol transport pathway. It can be reasonably deduced that the ginger, which exhibits antioxidant and anti-inflammatory properties, may prove beneficial in optimising this pathway. In light of the findings from experimental studies examining the effects of ginger-derived compounds on cholesterol efflux pathways, this study aims to investigate the impact of oral ginger supplementation on HDL function.

The crossover and double-blind study will be conducted in two four-week periods, with a washout period of at least three weeks between the two. The study population will be comprised of individuals who meet the following criteria: individuals between the ages of 18 and 75 years, with a body mass index less than 35 kg/m², who have not used serum lipid-lowering drugs in the previous month and have not regularly consumed ginger or ginger supplements (more than twice a week). In one of the two study periods, participants will ingest a ginger-based supplement in a dosage of 1500 mg, comprising three 500 mg capsules. In the other period, they will receive a placebo in the form of three capsules containing corn flour. A simple randomization method based on the RAS software is employed. To maintain the blind, the placebo and ginger capsules will be packed and coded in similar cans by an individual external to the study, and these capsules will remain sealed. At baseline and end of each study period, 6 cc of venous blood samples will be obtained from individuals after an overnight fast. The plasma and buffy coat (containing white blood cells) will be separated and stored at -80. Anthropometric measurements, including body weight, and blood pressure assessments will be conducted at baseline and end of each period. Additionally, a 24-hour food recall will be performed at both time points. The human monocyte cell line (THP-1) will be cultures in RPMI 1640 medium and subsequently differentiated into macrophage cells through the use of phorbol myristate acetate. Following differentiation, fluorescent cholesterol will be introduced to the culture medium in order to label the cells with this cholesterol. Subsequently, the plasma of the participants will be incorporated into the culture medium. Following the designated incubation period, the medium surrounding the cells will be removed and the cells will be lysed. The fluorescence of cholesterol in the medium and in the extract of THP-1 cells will be quantified using a fluorescence plate reader, allowing the calculation of CEC. The gene expression of ATP-binding cassette transporters A1 (ABCA1) and ATP-binding cassette transporters G1 (ABCG1) in the buffy coat obtained from blood samples of participants will be determined by quantitative polymerase chain reaction.

ELIGIBILITY:
Inclusion Criteria:

* a body mass index less than 35 kg/m², Exclusion Criteria:

Exclusion Criteria:

* Those with an allergy or sensitivity to ginger
* Those who have used serum lipid-lowering or antiinflammatory drugs in the previous month regularly
* Those who have regularly consumed ginger or ginger supplements (more than twice a week)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-11-03 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Ex-vivo plasma cholesterol efflux capacity | up to 6 weeks
  The ex vivo plasma cholesterol efflux capacity of THP-1 cells labeled with fluorescent cholesterol
Expression of ABCA1 and ABCG1 | up to 6 weeks
  The expression of genes encoding the ATP-binding cassette transporters ABCA1 and ABCG1 in peripheral white blood cells

SECONDARY OUTCOMES:
Plasma lipid profile | up to 6 weeks
  The plasma concentrations of triglycerides, cholesterol, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol
Plasma inflammatory biomarkers | up to 6 weeks
  The plasma concentrations of c-reactive protein, interleukin 6

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrition Clinic located in the Faculty of Nutrition Sciences, Shahid Beheshti University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided